CLINICAL TRIAL: NCT00439556
Title: Bortezomib (Velcade®) and Reduced-Intensity Allogeneic Stem Cell Transplantation for Patients With Lymphoid Malignancies
Brief Title: Bortezomib and Chemotherapy in Treating Participants With Lymphoid Malignancies Undergoing Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0066; NCI-2018-01830 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0066 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: CD20 Positive; Hematopoietic and Lymphoid Cell Neoplasm; Lymphocytic Neoplasm; Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma | interventions — Antilymphocyte Serum; thymoglobulin; Bortezomib; Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Melphalan; Methotrexate; merphos; Rituximab; CT-P10; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, transplant, filgrastim, tacrolimus) (Experimental): See Detailed Description
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Bortezomib; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Biological: Filgrastim; Drug: Melphalan; Drug: Methotrexate; Biological: Rituximab; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic stem cell transplantation
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase II trial studies the side effects and best dose of bortezomib when given with chemotherapy and to see how well they work in treating participants with lymphoid malignancies undergoing stem cell transplant. Giving chemotherapy before a stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the participant they may help the participant's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells called graft versus host disease. Giving tacrolimus and methotrexate after the transplant may stop this from happening. Giving bortezomib and chemotherapy may work better in treating participants with lymphoid malignancies undergoing a stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of Velcade (bortezomib) in patients with lymphoid malignancies undergoing allogeneic peripheral blood stem cell or bone marrow transplantation.

II. To determine the 1-year disease-free-survival (DFS) and the toxicity profile of Velcade (bortezomib) in patients with lymphoid malignancies undergoing allogeneic peripheral blood stem cell or bone marrow transplantation.

SECONDARY OBJECTIVES:

I. To compare the incidence of graft versus host disease (GVHD) with historical controls.

OUTLINE: This is a dose-escalation study of bortezomib.

Participants receive carmustine intravenously (IV) over 1 hour on day -6, cytarabine IV over 1 hour twice daily (BID) on days -5 to -2, etoposide IV over 3 hours BID on days -5 to -2, and melphalan IV over 30 minutes on day -1. Participants also receive rituximab IV on days -13, -6, +1, and +8, and bortezomib IV over 1 minute on days -13, -6, -1, and +2. Participants receiving a matched unrelated or mismatched donor transplant also receive anti-thymocyte globulin IV over 4-6 hours on days -6 and -5. Participants then undergo allogeneic hematopoietic stem cell transplantation over 30-45 minutes on day 0 and receive filgrastim subcutaneously (SC) once daily (QD) starting on day +7 until blood counts return to normal level. Participants receive tacrolimus IV starting on day -2 changing to orally (PO) before leaving the hospital for 6-8 months after the transplant. Participants also receive methotrexate IV over a few minutes on days +1, +3, and +6 and those receiving a matched unrelated or mismatched donor transplant also receive methotrexate IV on day +11.

After completion of study treatment, participants are followed up at 1 month, every 3 months for 1 year, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Any histological subtype of CD20+ lymphoid malignancies or T-cell lymphoid malignancies.
* Patients with CD20+ lymphoid malignancies in relapse after failing >= 1 prior regimen of conventional treatment and not eligible for non-myeloablative transplant. Patients with T-cell lymphoid malignancies can either be in relapse or newly diagnosed with high risk features (such as high International Prognostic Index [IPI] of >= 2).
* Patients with prior non-myeloablative transplant are eligible if not from the same donor.
* A fully-matched or one-antigen mismatched sibling or unrelated donor.
* Left ventricular ejection fraction (EF) >= 40% with no uncontrolled arrhythmias or symptomatic heart disease.
* Forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO) >= 40%.
* Serum creatinine < 1.8 mg/dL.
* Serum bilirubin < 3 X upper limit of normal.
* Serum glutamate pyruvate transaminase (SGPT) < 3 X upper limit of normal.
* Voluntary signed, written Institutional Review Board (IRB)-approved informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* Past history of anaphylaxis following exposure to rituximab or Velcade, boron or mannitol.
* History of grade 3 or 4 National Cancer Institute (NCI) toxicity with prior Velcade therapy.
* Patient with active central nervous system (CNS) disease.
* Pregnant (positive beta human chorionic gonadotropin [HCG] test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization) or currently breast feeding. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Known infection with human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV-I), hepatitis B, or hepatitis C.
* Patients with other malignancies diagnosed within 2 years prior to study day -13 (except skin squamous or basal cell carcinoma).
* Active uncontrolled bacterial, viral or fungal infections.
* Major surgical procedure or significant traumatic injury within 4 weeks prior to day -13.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 3 months prior to day -13.
* History of stroke within 6 months.
* Myocardial infarction within the past 6 months prior to study day 1, or has New York Heart Association (NYHA) class III or IV heart failure or arrhythmia, unstable angina, uncontrolled congestive heart failure or arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiography (ECG) abnormality at screening must be documented by investigator as not medically relevant.
* Uncontrolled hypertension (>= 140/90).
* Uncontrolled chronic diarrhea.
* A prior allogeneic transplant from the same donor.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has received other investigational drugs within 3 weeks before enrollment.
* Active peripheral neuropathy greater or equal to grade 2.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02-13 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa Khouri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled at MD Anderson clinic from February 2007 through May 2011.
Groups:
- Velcade Dose Level 1: BEAM (Carmustine/Etoposide/Cytarabine/Melphalan) + Rituxan + ATG (Thymoglobulin) (MUD pts only) + Velcade 1.0mg/m2 + ALLO SCT
- Velcade Dose Level 2: BEAM + Rituxan + ATG(MUD pts only) + Velcade 1.3mg/m2 + ALLO SCT
- Velcade Dose Level 3: BEAM + Rituxan + ATG(MUD pts only) + Velcade 1.6mg/m2 + ALLO SCT
Period: Overall Study
Arm/Group | Velcade Dose Level 1 | Velcade Dose Level 2 | Velcade Dose Level 3
Started | 36 | 4 | 0
Completed | 36 | 3 | 0
Not Completed | 0 | 1 | 0
Not completed — Patient was taken off study for non-comp | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients up to 70 years of age with any histological subtype of CD20+ lymphoid malignancy or T-Cell lymphoid malignancy who were not eligible for a non-myeloablative transplant.
Groups:
- Velcade Dose Level 1: BEAM + Rituxan + ATG(MUD pts only) + Velcade (1-1.3mg/m2) + ALLO SCT
- Total: Total of all reporting groups
Arm/Group | Velcade Dose Level 1 | Velcade Dose Level 2 | Velcade Dose Level 3 | Total
Number analyzed (Participants) | 36 | 3 | 0 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 3 | 0 | 39
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 54 [22 to 65] | 58 [47 to 65] |  | 54 [22 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 |  | 9
  Male | 28 | 2 |  | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 |  | 5
  Not Hispanic or Latino | 4 | 0 |  | 4
  Unknown or Not Reported | 27 | 3 |  | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 2 | 0 |  | 2
  White | 32 | 3 |  | 35
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 2 | 0 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 3 |  | 39
Breakdown of Disease by Number of Participants in each Dose Level [Count of Participants; unit: Participants] — Patients up to 70 years of age with any histological subtype of CD20+ lymphoid malignancy or T-Cell lymphoid malignancy who were not eligible for a non-myeloablative transplant.
  Participants
    Large Cell Lymphoma | 9 | 2 |  | 11
    CLL | 12 | 1 |  | 13
    Folicular Lymphoma | 8 | 0 |  | 8
    Mantle Cell Lymphoma | 2 | 0 |  | 2
    Marginal Zone Lymphoma | 1 | 0 |  | 1
    T-Cell Lymphoma | 4 | 0 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: To determine the maximum tolerated dose(MTD) of velcade and dose limiting toxicity(DLT). A dose limiting toxicity (DLT) was defined as a grade 3-4 neurological toxicity, graft failure, or death due to GvHD. The Commom Terminlogy Criteria for Adverse Events v3.0 was used.
Time Frame: From start of treatment to 90 days after the start of treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy, Transplant, Filgrastim, Tacrolimus): BEAM + Rituxan + ATG(MUD pts only) + Velcade (1-1.3mg/m2) + ALLO SCT
Arm/Group | Treatment (Chemotherapy, Transplant, Filgrastim, Tacrolimus) | Velcade Dose Level 2 | Velcade Dose Level 3
Number analyzed (Participants) | 36 | 3 | 0
Participants | 0 | 0 | 0

2. Primary Outcome: Disease-free Survival
Description: To determine DFS at 1 year post transplant.
Time Frame: At 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Velcade Dose Level 1: BEAM + Rituxan + ATG(MUD pts only) + Velcade 1.0mg/m2 + ALLO SCT
Arm/Group | Velcade Dose Level 1 | Velcade Dose Level 2 | Velcade Dose Level 3
Number analyzed (Participants) | 36 | 3 | 0
Participants | 16 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 100 Days post transplant
Description: There were no participants enrolled on Velcade dose level 3
Groups:
- Gemcitabine Dose Level 3: BEAM + Rituxan + ATG(MUD pts only) + Velcade 1.6mg/m2 + ALLO SCT
Arm/Group | Velcade Dose Level 1 | Velcade Dose Level 2 | Gemcitabine Dose Level 3
All-Cause Mortality (participants affected / at risk) | 6/36 | 2/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 6/36 | 2/3 | 0/0
Other Adverse Events (participants affected / at risk) | 36/36 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade Dose Level 1 (N=36) | Velcade Dose Level 2 (N=3) | Gemcitabine Dose Level 3 (N=0)
Infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Acute GvHD(graft vs Host Disease) (General disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade Dose Level 1 (N=36) | Velcade Dose Level 2 (N=3) | Gemcitabine Dose Level 3 (N=0)
Dysrhythmia (Cardiac disorders) | 4 (4) | 0 (0) | NA
Decreased Cardiac Function (Cardiac disorders) | 3 (3) | 0 (0) | NA
Hypertension (Cardiac disorders) | 5 (5) | 0 (0) | NA
Fluid Overload (General disorders) | 13 (13) | 3 (3) | NA
Fever (General disorders) | 13 (14) | 0 (0) | NA
Diarrhea (Gastrointestinal disorders) | 23 (23) | 3 (3) | NA
Mucositis (Gastrointestinal disorders) | 12 (12) | 2 (2) | NA
Nausea (Gastrointestinal disorders) | 31 (31) | 3 (3) | NA
Elevated Creatinine (Renal and urinary disorders) | 3 (3) | 2 (2) | NA
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1) | NA
Transaminitis (Hepatobiliary disorders) | 5 (5) | 0 (0) | NA
Infection (Infections and infestations) | 27 (56) | 3 (5) | NA
Neutropenic Fever (Infections and infestations) | 19 (19) | 0 (0) | NA
SOB (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | NA
Acute GvHD (General disorders) | 24 (41) | 1 (1) | NA
Chronic GvHD (General disorders) | 7 (9) | 2 (2) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT00439556/Prot_SAP_000.pdf